CLINICAL TRIAL: NCT00798382
Title: Comparative Gastrointestinal Tolerance of Various Infant Formulas in Healthy Term Infants
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Abbott Nutrition (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AK54
Record Dates: First submitted 2008-11-25; First posted 2008-11-26 (Estimated); Last update posted 2012-06-14 (Estimated); Status verified 2012-06

CONDITIONS: Infant, Newborn

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1: Soy formula (Experimental): experimental soy formula #1
  Interventions: Other: soy protein formula
- 2: Soy Formula (Active Comparator): Commercially available soy formula
  Interventions: Other: Commercially available soy formula
- 3: Soy formula (Experimental): experimental soy formula #2
  Interventions: Other: Soy formula experimental #2

INTERVENTIONS:
Other: soy protein formula — ad lib for 0-35 days of age
  Other Names: experimental soy formula
  Arms: 1: Soy formula
Other: Commercially available soy formula — ad lib for 0-35 days of age
  Arms: 2: Soy Formula
Other: Soy formula experimental #2 — ad lib for 0-35 days of age
  Other Names: Experimental soy formula
  Arms: 3: Soy formula

SUMMARY:
The objective of this study is to assess the comparative gastrointestinal (GI) tolerance of normal term infants to two experimental soy-based formulas, relative to a commercially available soy-based formula.

ELIGIBILITY:
Inclusion Criteria:

* Infant is judged to be in good health.
* Infant is a singleton from a full term birth with a gestational age of 37-42 weeks.
* Infant's birth weight was > 2490 g (~5 lb 8 oz).
* Infant is between 0 and 8 days of age at enrollment.
* Parent(s) confirm their intention to feed their infant the study product as the sole source of nutrition for the duration of the study.
* Parent(s) confirm their intention not to administer vitamin or mineral supplements, solid foods or juices to their infant for the duration of the study.
* Infants using medications or home remedies, herbal preparations or rehydration/intravenous (IV) fluids that might affect GI tolerance may not be enrolled.

Exclusion Criteria:

* An adverse maternal, fetal or infant medical history that is thought by the investigator to have potential for effects on tolerance, growth, and/or development.
* Infant has been treated with antibiotics.
* Infant has received probiotics.

Max Age: 8 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 154 (Actual)
Dates: Start 2008-12; Primary Completion 2009-04 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Gastrointestinal tolerance from Study Visit 1 to Study Visit 3 at 35 days of age. | 35 days

SECONDARY OUTCOMES:
Additional gastrointestinal measures of tolerance from Study Visit 1 to Study Visit 3 at 35 days of age | 35 days

CONTACTS AND LOCATIONS:
Overall Officials: John Lasekan, PhD, Study Chair — Abbott Nutrition
Locations (17):
- United States (17):
  - Arkansas Children's Hospital Research Institute, Little Rock, Arkansas
  - All Women's Heatlthcare of West Broward, Inc: Discovery Clinical Research, Inc, Plantation, Florida
  - SCORE Physician Alliance, LLC, St. Petersburg, Florida
  - University of South Florida Health Pediatrics, Tampa, Florida
  - North Georgia Clinical Research, Dalton, Georgia
  - Medical Associates Clinic, Dubuque, Iowa
  - Kentucky Pediatric Research, Bardstown, Kentucky
  - PediaResearch, LLC, Owensboro, Kentucky
  - Midwest Children's Health Research Institute, LLC, Lincoln, Nebraska
  - Center for Human Nutrition, Omaha, Nebraska
  - Pediatric Associates of Mount Carmel, Inc, Cincinnati, Ohio
  - MetroHealth Medical Center, Cleveland, Ohio
  - Dayton Clinical Research, Dayton, Ohio
  - Ohio Pediatric Research Association, Huber Heights, Ohio
  - Institute of Clinical Research, LLC, Mayfield Heights, Ohio
  - Primary Physician's Research, Inc, Pittsburgh, Pennsylvania
  - West Virginia University, Department of Pediatrics, Morgantown, West Virginia